CLINICAL TRIAL: NCT03253913
Title: Resveratrol and Sirolimus in Lymphangioleiomyomatosis Trial (RESULT)
Brief Title: Resveratrol and Sirolimus in Lymphangioleiomyomatosis Trial
Acronym: RESULT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nishant Gupta, MD, MS, Adjunct Assistant Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-4904; 1R34HL138235-01 (NIH)
Record Dates: First submitted 2017-08-10; First posted 2017-08-18 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Sirolimus; Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Resveratrol 250mg daily for the first 8 weeks, followed by 250mg twice daily for the next 8 weeks, and then 500mg twice daily for the last 8 weeks.
  Patients will be on a stable background therapy of sirolimus prior to enrolling and will continue on that regimen throughout the study.
  Interventions: Drug: Sirolimus; Drug: Resveratrol

INTERVENTIONS:
Drug: Sirolimus — Patients will have been on a stable dose of sirolimus prior to enrolling and will continue that throughout the study.
  Other Names: Rapamycin
Drug: Resveratrol — Escalating doses of resveratrol will be given throughout the study. Patients will start at 250mg daily for 8 weeks, followed by 500mg daily for 8 weeks, and 500mg BID for the last 8 weeks.

SUMMARY:
RESULT is a phase II dose-escalating, open-label, safety and efficacy study to determine if there is a potential benefit of resveratrol in combination with sirolimus in patients with lymphangioleiomyomatosis (LAM). The primary study objective is to assess the change in serum vascular endothelial growth factor-D (VEGF-D) level after 24 weeks of treatment with a combination of resveratrol and sirolimus as compared to the VEGF-D level in patients on a stable dose of sirolimus alone. The secondary objectives of this study include an assessment of the safety and adverse effect profile of combined resveratrol and sirolimus in adult patients with LAM, and to determine the effect of treatment with a combination of resveratrol and sirolimus on changes in lung function and quality of life.

DETAILED DESCRIPTION:
Study Design RESULT was an open label, dose-escalation, phase 2 study with longitudinal repeated measures. In order to be eligible for trial inclusion, patients had to satisfy all of the following criteria: 1) confirmed diagnosis of LAM per the American Thoracic Society/Japanese Respiratory Society Clinical Practice Guidelines14, 2) age ≥18 years with signed informed consent, 3) on sirolimus for at least 20 weeks, and 4) VEGF-D stabilization as demonstrated by two stable values post initiation of sirolimus and drawn at least 12 weeks apart from each other. Key exclusion criteria included inability to provide consent, active listing for lung transplantation, enrolled in another interventional clinical trial, known allergy or hypersensitivity to resveratrol, and current or planned pregnancy in the next six months.

RESULT was a single site study conducted at the University of Cincinnati (UC). Study enrollment was open to LAM patients throughout the United States with travel reimbursement provided through the study. The study was reviewed and approved by UC's Institutional Review Board (IRB 2016-4904). An independent Data and Safety Monitoring Board (DSMB) was convened and met every six months to ensure the safety of study participants. All subjects provided written informed consent prior to the conduct of any study related activity.

Outcome Measures The primary objective of this study was to assess the change in serum VEGF-D value after 24 weeks of treatment with a combination of resveratrol and sirolimus, as compared to the historical VEGF-D values of patients prior to the study on sirolimus alone. Serial assessments of serum VEGF-D, pulmonary function tests (PFTs), treatment related adverse effects (AEs), complete blood count, liver and renal function tests, and HRQOL were performed at baseline and at 8, 16, and 24 weeks. In addition, sirolimus trough levels, measured 24 +/- 4 hours following the last dose, were assessed at baseline and at weeks 2, 4, 8, 12, 16, 18, 20 and 24. VEGF-D quantification was performed at the Translational Trial Development and Support Laboratory based at Cincinnati Children's Hospital Medical Center in a College of American Pathologists (CAP)/Clinical Laboratory Improvement Amendments (CLIA) approved manner. All other laboratory assessments were performed via Quest Diagnostics. HRQOL was measured by using four validated scales: St. George's Respiratory Questionnaire (SGRQ), University of California San Diego Shortness of Breath score (SDSOB), EuroQol visual analogue scale (EQVAS), and A Tool to Assess Quality of Life in LAM (ATAQ-LAM).

Study Drug Resveratrol used in this study was obtained from Evolva and manufactured by fermentation using genetically modified yeast in a process that results in trans-resveratrol with a purity of at least 98%, and packaged into capsules with each capsule containing 125mg resveratrol. The capsules were independently verified for content by mass spectrometry performed at UC and for sterility by microbial testing at Q Laboratories Inc., Cincinnati. Investigational new drug (IND) designation for studying Resveratrol in this trial was obtained from the United States Food and Drug Administration (FDA): IND 131722; IND Sponsor: N. Gupta.

Resveratrol was administered in a stepwise dose escalating fashion at 8-week intervals with assessment of VEGF-D, PFTs, AEs, and HRQOL prior to each dose escalation. The starting dose of resveratrol was 250mg once daily for the first 8 weeks, followed by 500mg daily from Weeks 8 - 16, and 500mg twice daily for the last 8 weeks (Weeks 16 - 24), with provisions for dose reduction if necessitated by AEs. Treatment related AEs were tabulated using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the trial must meet all of the following criteria.

1. Definitive diagnosis LAM based on the presence of characteristic cystic change on high-resolution computed tomography (HRCT) of the chest. The diagnosis must be confirmed by one of the following:

   A) Histopathological confirmation by biopsy (lung, abdominal mass, lymph node or kidney or cytology from thoracic or abdominal sources revealing human melanoma black-45 (HMB45)+ staining of spindled/epithelioid cells) B) Compatible chest CT scan findings in the setting of tuberous sclerosis, angiomyolipomas (diagnosed by CT, magnetic resonance imaging (MRI) by the site radiologist or biopsy) or chylous pleural effusion (verified by tap) C) Chest CT scan findings compatible with LAM and a VEGF-D level ≥ 800pg/ml.
2. Age 18 years or greater.
3. Signed and dated informed consent
4. Currently on sirolimus for treatment of LAM for at least 20 weeks
5. Evidence of disease stabilization on sirolimus as demonstrated by two stable values of serum VEGF-D post initiation of sirolimus drawn at least 12 weeks apart from each other. For the purpose of this study, a variation in serum VEGF-D of less than or equal to 15% is considered stable.

Exclusion Criteria:

* Subjects who meet any of the following criteria are not eligible for enrollment as study participants:

  1. Known allergy or hypersensitivity to Resveratrol
  2. Inability to provide informed consent
  3. Active enrollment in other clinical drug trials for LAM
  4. Pregnant or plan to become pregnant in the next 6 months
  5. Breast feeding
  6. Inability to comply with pulmonary function tests or follow up visits
  7. Inadequate contraception
  8. Use of estrogen containing medications within the 30 days prior to randomization
  9. History of organ transplant
  10. Actively listed for lung transplantation
  11. Inability to comply with study procedures or attend scheduled study visits
  12. Any clinically significant medical disease (other than LAM) that is associated with an expected survival of less than 2 years, or likely to impact the ability of the patient to participate in the study in the opinion of the investigator, or impact the study efficacy or safety assessments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — LAM is a disease that almost exclusively involves females. Thus trial participants will be females only.
Enrollment: 25 (Actual)
Dates: Start 2018-03-31 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nishant Gupta, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gupta N, Zhang B, Zhou Y, McCormack FX, Ingledue R, Robbins N, Kopras EJ, McMahan S, Singla A, Swigris J, Cole AG, Holz MK. Safety and Efficacy of Combined Resveratrol and Sirolimus in Lymphangioleiomyomatosis. Chest. 2023 May;163(5):1144-1155. doi: 10.1016/j.chest.2023.01.007. Epub 2023 Jan 13. PMID 36642366

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Resveratrol 250mg daily for the first 8 weeks, followed by 250mg twice daily for the next 8 weeks, and then 500mg twice daily for the last 8 weeks.
  Patients will be on a stable background therapy of sirolimus prior to enrolling and will continue on that regimen throughout the study.
  Sirolimus: Patients will be on a stable dose of sirolimus prior to enrolling and will continue that throughout the study.
  Resveratrol: Escalating doses of resveratrol will be given throughout the study. Patients will start at 250mg daily for 8 weeks, followed by 500mg daily for 8 weeks, and 500mg BID for the last 8 weeks.
Period: First 8 Weeks (250mg Daily Resveratrol)
Arm/Group | Treatment Arm
Started | 25
Completed | 25
Not Completed | 0
Period: Weeks 8 - 16 (Resveratrol 500mg Daily)
Arm/Group | Treatment Arm
Started | 25
Completed | 25
Not Completed | 0
Period: Weeks 16-24 (Resveratrol 1,000mg Daily)
Arm/Group | Treatment Arm
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [47 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Serum Vascular Endothelial Growth Factor-D (VEGF-D) Levels After Treatment With a Combination of Resveratrol and Sirolimus as Compared to Baseline Serum VEGF-D Levels on Sirolimus Alone
Description: Change in serum VEGF-D level in pg/ml after treatment with a combination of resveratrol and sirolimus as compared to the historical VEGF-D level in patients on a stable dose of sirolimus alone. Baseline VEGF-D values represent serum VEGF-D levels on stable dose of sirolimus alone prior to starting study drug.
Time Frame: Baseline, Week 8, Week 16, Week 24
Population: Longitudinal slope of serum VEGF-D levels
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
pg/ml
  Baseline VEGF-D level in patients on a stable dose of sirolimus alone | 617 [489 to 677]
  Week 8 | 543 [455 to 704]
  Week 16 | 581 [485 to 724]
  Week 24 | 575 [448 to 673]

2. Secondary Outcome: Number of Treatment-Emergent Adverse Events
Description: Safety and adverse effect profile of combined resveratrol and sirolimus in adult patients with LAM
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Number; unit: Adverse effects
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
Adverse effects
  250 mg daily | 42
  500mg daily | 25
  1000mg daily | 25

3. Secondary Outcome: Change in Forced Expiratory Volume in One-second (FEV1) After 24 Weeks of Combined Treatment With Resveratrol and Sirolimus
Description: Difference in the absolute Forced expiratory volume in one-second (FEV1) after 24 weeks of treatment. FEV1 values reported are in liters. There are no definite minimum and maximum values of FEV1 as it is a physiological measure of lung function and varies from individual to individual. Higher FEV1 scores indicate better lung function.
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Median (Inter-Quartile Range); unit: Absolute FEV1 in liters
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
Absolute FEV1 in liters
  Baseline | 1.74 [1.46 to 2.3]
  Week 8 | 1.98 [1.4 to 2.36]
  Week 16 | 2.01 [1.18 to 2.57]
  Week 24 | 1.94 [1.2 to 2.59]

4. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Quality of Life Assessment Scores After Treatment With Combined Resveratrol and Sirolimus
Description: Quality of life scores will be calculated by using SGRQ to determine if the combination of resveratrol and sirolimus can improve the quality of life in patients with LAM. This is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating worse quality of life.
Time Frame: Baseline, Week 8, Week 16, Week 24.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
score on a scale
  Baseline | 42 [39 to 46]
  Week 8 | 43.5 [38 to 49]
  Week 16 | 43 [40 to 49]
  Week 24 | 42 [39 to 47]

5. Secondary Outcome: Scores on "A Tool to Assess Quality of Life in LAM (ATAQ-LAM) Quality of Life Assessment" Scale After Treatment With 24 Weeks of Resveratrol and Sirolimus
Description: Quality of life scores will be calculated by using ATAQ-LAM to determine if the combination of resveratrol and sirolimus can improve the quality of life in patients with LAM. A Tool to Assess Quality of Life in LAM (ATAQ-LAM) is a disease-specific instrument designed to assess HRQOL in patients with LAM, and consists of 32 items divided into 4 domains: exertional dyspnea, cough, fatigue, and emotional well-being. The total scores on this scale can range between 32 - 192, with higher scores indicating worse quality of life.
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
score on a scale
  Baseline | 72 [54 to 88]
  Week 8 | 70 [49 to 101]
  Week 16 | 60 [44 to 82]
  Week 24 | 57 [47 to 87]

6. Secondary Outcome: San Diego Shortness of Breath Score (SD-SOB) Quality of Life Assessment Scores After Treatment With 24 Weeks of Resveratrol and Sirolimus
Description: The San Diego shortness of breath questionnaire measures the quality-of-life impairment secondary to dyspnea resulting from pulmonary disorders. It is a 24-item measure that assesses self-reported shortness of breath while performing a variety of activities of daily living, with higher scores indicating worse quality of life.
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
score on a scale
  Baseline | 29 [21 to 35]
  Week 8 | 31 [16 to 44]
  Week 16 | 23 [15 to 42]
  Week 24 | 22 [12 to 40]

7. Secondary Outcome: EuroQOL Visual Analogue Scale (EQ-5D) Scores After Treatment With 24 Weeks of Sirolimus and Resveratrol.
Description: The EuroQOL visual-analogue scale (EQVAS) measures self-reported ratings of health status. Scores range from 0 to100, with lower scores indicating worse functioning.
Time Frame: Baseline, Week 8, Week 16, Week 24
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 25
score on a scale
  Baseline | 80 [65 to 85]
  Week 8 | 85 [75 to 90]
  Week 16 | 90 [75 to 95]
  Week 24 | 90 [80 to 90]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse effects were tabulated using the National Cancer Institute's Common Terminology Criteria for Adverse Events version 4.
Groups:
- 250mg Resveratrol Daily (First 8 Weeks): 250mg resveratrol added to pre-existing sirolimus
- 500mg Daily Resveratrol (Weeks 8 - 16): 500mg resveratrol added to pre-existing sirolimus
- 1,000mg Daily Resveratrol: 1,000mg resveratrol added to pre-existing sirolimus
Arm/Group | 250mg Resveratrol Daily (First 8 Weeks) | 500mg Daily Resveratrol (Weeks 8 - 16) | 1,000mg Daily Resveratrol
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 14/25 | 5/25 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250mg Resveratrol Daily (First 8 Weeks) (N=25) | 500mg Daily Resveratrol (Weeks 8 - 16) (N=25) | 1,000mg Daily Resveratrol (N=25)
nausea (Gastrointestinal disorders) | 3 (4) | 2 (2) | 2 (3)
diarrhea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
gastrointestinal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (4)
Infection (Infections and infestations) | 6 (7) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT03253913/Prot_SAP_001.pdf